CLINICAL TRIAL: NCT06467383
Title: A Study to Describe the Diagnostic and Therapeutic Path of Patients with NSCLC in Early Stage and Locally Advanced
Acronym: Key-Early
Status: Recruiting | Type: Observational
Sponsor: MSD Italia S.r.l. (Industry)
Collaborators: YGHEA, CRO Division of Ecol Studio spa (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS009903
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer; NSCLC; NSCLC, Stage III; NSCLC, Stage I
Keywords: NSCLC early stage; NSCLC locally advanced; retrospective observational study; Real-World Evidence
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a non-interventional, retrospective observational study to improve knowledge regarding the diagnosis and treatments of patients who have/had non-small cell lung cancer (NSCLC), either early stage (stage I-II).

DETAILED DESCRIPTION:
Due to heterogeneity of patients with stage I-III Non Small Cell Lung Cancer (NSCLC), there is not a unique common therapeutic approach and there is no consensus about the optimal timing, sequencing and combination of surgery, chemotherapy and radiotherapy across the spectrum of early stage and locally advance disease. Consequently, the choice of local treatment modality can vary across countries and centers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage I-III NSCLC who have received curative surgery or radiotherapy between January 2018 and June 2019 with available follow-up through January 2021
2. Adult patients (aged ≥ 18 years) at the moment of diagnosis
3. Patients (or their legally acceptable representatives) must have signed and dated the Informed Consent form; privacy Form (ICF). In case of deceased or untraceable patient the investigator before collecting data shall demonstrate and report all necessary measures adopted to contact the patient.

Exclusion Criteria:

1. Patients without availability of medical charts or information required
2. Enrollment in studies imposing a specific patient's management strategy which does not correspond to the site's normal clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with early stage and locally advanced NSCLC (stage I-III) who had completed curative treatment planning and subsequent at least 18-months follow-up between January 2018 and January 2021.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-24 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
NSCLC treatment approaches in Real-World practice | Restrospective data capture from January 2018 to January 2021.
  Percentage of patients undergoing to:
  1. surgical resection of the lung cancer with curative intent;
  2. definitive (chemo)radiotherapy (defined as any regimen of chemotherapy administered with concurrent radiotherapy)
  3. neoadjuvant treatment (4 cycles) before surgery
  4. adjuvant treatments (4 cycles) after surgery
Percentage of patients discusses in multidisciplinary team | Restrospective data capture from January 2018 to January 2021
  Multidisciplinary team defined as the involvement of radiotherapy unit, pneumology and/or interventional pneumology unit in patient discussion.
Healthcare resource utilization aof different therapeutic approaches | Restrospective data capture from January 2018 to January 2021.
  Healthcare resources used to manage the patients will be described in terms of lab tests and/or outpatient visits and/or drug therapy and/or diagnostic tests.
Direct medical costs of different therapeutic approaches | Restrospective data capture from January 2018 to January 2021.
  The cost of the therapeutic approach (cost of illness) will be estimated through an activity-based costing (ABC) technique which allows to calculate the full cost of a service by measuring the cost of each individual activity/resource related to it.

SECONDARY OUTCOMES:
NSCLC treatments timeline in Real-World practice | Restrospective data capture from January 2018 to January 2021.
  Median Time from:
  1. diagnosis/multidisciplinary referral to surgery or start of radioterapy
  2. surgery/completion of Radiotherapy to satrt of adjiuvant treatmen

OTHER OUTCOMES:
Biomarkers profile evaluation at NSCLC diagnosis | Restrospective data capture from January 2018 to January 2021.
  Percentage of PD-L1, EGFR/ALK, KRAS test performed along with results
PD-L1 Biomarker profile evaluation at NSCLC diagnosis | Restrospective data capture from January 2018 to January 2021.
  Percentage of PD-L1 test performed along with results
EGFR/ALK Biomarkers profile evaluation at NSCLC diagnosis | Restrospective data capture from January 2018 to January 2021.
  Percentage of EGFR/ALK test performed along with results
KRAS Biomarkers profile evaluation at NSCLC diagnosis | Restrospective data capture from January 2018 to January 2021.
  Percentage of KRAS test performed along with result

CONTACTS AND LOCATIONS:
Overall Officials: Giada Iuliano, MD, Study Chair — MSD Italia srl
Locations (25):
- Italy (25):
  - IRCCS Casa di sollievo dalla sofferenza, San Giovanni Rotondo, FG
  - ASST degli Spedali Civili di Brescia, Brescia
  - Gemelli Molise, Campobasso
  - Humanitas Istituto Clinico Catanese, Catania
  - Policlinico Rodolico, Catania
  - AOU Careggi, Florence
  - IRCCS Policlinico S. Martino, Genova
  - AO Papardo, Messina
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Clinico Humanitas, Milan
  - Istituto Nazionale dei Tumori - Fondazione IRCCS, Milan
  - AOU dei Colli - Monaldi, Napoli
  - AOU Vanvitelli, Napoli
  - A.O.U. Maggiore della Carità di Novara, Novara
  - IOV - Istituto Oncologico veneto - IRCCS, Padua
  - AOUP Policlinico Giaccone, Palermo
  - Azienda Ospedaliera Perugia - Ospedale S. Maria della MIsericordia, Perugia
  - Azienda USL Toscana Centro - Ospedale san Jacopo, Pistoia
  - Centro di Riferimento Oncologico IRCCS, Pordenone
  - Azienda Ospedaliera Regionale San Carlo di Potenza, Potenza
  - AUSL Romagna Ospedale Santa Maria delle Croci Ravenna, Ravenna
  - IRCCS AUSL Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario "A. Gemelli", Roma
  - ASST dei Sette Laghi, Varese
  - AOUI Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Postmus PE, Kerr KM, Oudkerk M, Senan S, Waller DA, Vansteenkiste J, Escriu C, Peters S; ESMO Guidelines Committee. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv1-iv21. doi: 10.1093/annonc/mdx222. No abstract available. PMID 28881918
- [Background] Rosen JE, Keshava HB, Yao X, Kim AW, Detterbeck FC, Boffa DJ. The Natural History of Operable Non-Small Cell Lung Cancer in the National Cancer Database. Ann Thorac Surg. 2016 May;101(5):1850-5. doi: 10.1016/j.athoracsur.2016.01.077. Epub 2016 Apr 1. PMID 27041452
- [Background] Jin G, Wang X, Xu C, Sun J, Yuan Z, Wang J, Zhao L. Disparities in survival following surgery among patients with different histological types of N2-III non-small cell lung cancer: a Surveillance, Epidemiology and End Results (SEER) database analysis. Ann Transl Med. 2020 Oct;8(20):1288. doi: 10.21037/atm-20-4357. PMID 33209868
- [Background] Ball D, Mai GT, Vinod S, Babington S, Ruben J, Kron T, Chesson B, Herschtal A, Vanevski M, Rezo A, Elder C, Skala M, Wirth A, Wheeler G, Lim A, Shaw M, Schofield P, Irving L, Solomon B; TROG 09.02 CHISEL investigators. Stereotactic ablative radiotherapy versus standard radiotherapy in stage 1 non-small-cell lung cancer (TROG 09.02 CHISEL): a phase 3, open-label, randomised controlled trial. Lancet Oncol. 2019 Apr;20(4):494-503. doi: 10.1016/S1470-2045(18)30896-9. Epub 2019 Feb 12. PMID 30770291
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Background] Senan S, Brade A, Wang LH, Vansteenkiste J, Dakhil S, Biesma B, Martinez Aguillo M, Aerts J, Govindan R, Rubio-Viqueira B, Lewanski C, Gandara D, Choy H, Mok T, Hossain A, Iscoe N, Treat J, Koustenis A, San Antonio B, Chouaki N, Vokes E. PROCLAIM: Randomized Phase III Trial of Pemetrexed-Cisplatin or Etoposide-Cisplatin Plus Thoracic Radiation Therapy Followed by Consolidation Chemotherapy in Locally Advanced Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Mar 20;34(9):953-62. doi: 10.1200/JCO.2015.64.8824. Epub 2016 Jan 25. PMID 26811519
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Benitez-Majano S, Fowler H, Maringe C, Di Girolamo C, Rachet B. Deriving stage at diagnosis from multiple population-based sources: colorectal and lung cancer in England. Br J Cancer. 2016 Jul 26;115(3):391-400. doi: 10.1038/bjc.2016.177. Epub 2016 Jun 21. PMID 27328310
- [Background] Blackstock AW, Govindan R. Definitive chemoradiation for the treatment of locally advanced non small-cell lung cancer. J Clin Oncol. 2007 Sep 10;25(26):4146-52. doi: 10.1200/JCO.2007.12.6581. PMID 17827465
- [Background] NSCLC Meta-analyses Collaborative Group; Arriagada R, Auperin A, Burdett S, Higgins JP, Johnson DH, Le Chevalier T, Le Pechoux C, Parmar MK, Pignon JP, Souhami RL, Stephens RJ, Stewart LA, Tierney JF, Tribodet H, van Meerbeeck J. Adjuvant chemotherapy, with or without postoperative radiotherapy, in operable non-small-cell lung cancer: two meta-analyses of individual patient data. Lancet. 2010 Apr 10;375(9722):1267-77. doi: 10.1016/S0140-6736(10)60059-1. Epub 2010 Mar 24. PMID 20338627
- [Background] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Background] Salazar MC, Rosen JE, Wang Z, Arnold BN, Thomas DC, Herbst RS, Kim AW, Detterbeck FC, Blasberg JD, Boffa DJ. Association of Delayed Adjuvant Chemotherapy With Survival After Lung Cancer Surgery. JAMA Oncol. 2017 May 1;3(5):610-619. doi: 10.1001/jamaoncol.2016.5829. PMID 28056112
- [Background] Artal Cortes A, Calera Urquizu L, Hernando Cubero J. Adjuvant chemotherapy in non-small cell lung cancer: state-of-the-art. Transl Lung Cancer Res. 2015 Apr;4(2):191-7. doi: 10.3978/j.issn.2218-6751.2014.06.01. PMID 25870801
- [Background] Pisters KM, Vallieres E, Crowley JJ, Franklin WA, Bunn PA Jr, Ginsberg RJ, Putnam JB Jr, Chansky K, Gandara D. Surgery with or without preoperative paclitaxel and carboplatin in early-stage non-small-cell lung cancer: Southwest Oncology Group Trial S9900, an intergroup, randomized, phase III trial. J Clin Oncol. 2010 Apr 10;28(11):1843-9. doi: 10.1200/JCO.2009.26.1685. Epub 2010 Mar 15. PMID 20231678
- [Background] Scagliotti GV, Pastorino U, Vansteenkiste JF, Spaggiari L, Facciolo F, Orlowski TM, Maiorino L, Hetzel M, Leschinger M, Visseren-Grul C, Torri V. Randomized phase III study of surgery alone or surgery plus preoperative cisplatin and gemcitabine in stages IB to IIIA non-small-cell lung cancer. J Clin Oncol. 2012 Jan 10;30(2):172-8. doi: 10.1200/JCO.2010.33.7089. Epub 2011 Nov 28. PMID 22124104
- [Background] Song WA, Zhou NK, Wang W, Chu XY, Liang CY, Tian XD, Guo JT, Liu X, Liu Y, Dai WM. Survival benefit of neoadjuvant chemotherapy in non-small cell lung cancer: an updated meta-analysis of 13 randomized control trials. J Thorac Oncol. 2010 Apr;5(4):510-6. doi: 10.1097/JTO.0b013e3181cd3345. PMID 20107424
- [Background] Felip E, Rosell R, Maestre JA, Rodriguez-Paniagua JM, Moran T, Astudillo J, Alonso G, Borro JM, Gonzalez-Larriba JL, Torres A, Camps C, Guijarro R, Isla D, Aguilo R, Alberola V, Padilla J, Sanchez-Palencia A, Sanchez JJ, Hermosilla E, Massuti B; Spanish Lung Cancer Group. Preoperative chemotherapy plus surgery versus surgery plus adjuvant chemotherapy versus surgery alone in early-stage non-small-cell lung cancer. J Clin Oncol. 2010 Jul 1;28(19):3138-45. doi: 10.1200/JCO.2009.27.6204. Epub 2010 Jun 1. PMID 20516435
- [Background] NSCLC Meta-analysis Collaborative Group. Preoperative chemotherapy for non-small-cell lung cancer: a systematic review and meta-analysis of individual participant data. Lancet. 2014 May 3;383(9928):1561-71. doi: 10.1016/S0140-6736(13)62159-5. Epub 2014 Feb 25. PMID 24576776
- [Background] Gilligan D, Nicolson M, Smith I, Groen H, Dalesio O, Goldstraw P, Hatton M, Hopwood P, Manegold C, Schramel F, Smit H, van Meerbeeck J, Nankivell M, Parmar M, Pugh C, Stephens R. Preoperative chemotherapy in patients with resectable non-small cell lung cancer: results of the MRC LU22/NVALT 2/EORTC 08012 multicentre randomised trial and update of systematic review. Lancet. 2007 Jun 9;369(9577):1929-37. doi: 10.1016/S0140-6736(07)60714-4. PMID 17544497
- [Background] Postoperative radiotherapy in non-small-cell lung cancer: systematic review and meta-analysis of individual patient data from nine randomised controlled trials. PORT Meta-analysis Trialists Group. Lancet. 1998 Jul 25;352(9124):257-63. PMID 9690404
- [Background] Douillard JY, Rosell R, De Lena M, Riggi M, Hurteloup P, Mahe MA; Adjuvant Navelbine International Trialist Association. Impact of postoperative radiation therapy on survival in patients with complete resection and stage I, II, or IIIA non-small-cell lung cancer treated with adjuvant chemotherapy: the adjuvant Navelbine International Trialist Association (ANITA) Randomized Trial. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):695-701. doi: 10.1016/j.ijrobp.2008.01.044. Epub 2008 Apr 24. PMID 18439766
- [Background] Mikell JL, Gillespie TW, Hall WA, Nickleach DC, Liu Y, Lipscomb J, Ramalingam SS, Rajpara RS, Force SD, Fernandez FG, Owonikoko TK, Pillai RN, Khuri FR, Curran WJ, Higgins KA. Postoperative radiotherapy is associated with better survival in non-small cell lung cancer with involved N2 lymph nodes: results of an analysis of the National Cancer Data Base. J Thorac Oncol. 2015 Mar;10(3):462-71. doi: 10.1097/JTO.0000000000000411. PMID 25384064
- [Background] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Gray JE, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, Cho BC, Planchard D, Paz-Ares L, Faivre-Finn C, Vansteenkiste JF, Spigel DR, Wadsworth C, Taboada M, Dennis PA, Ozguroglu M, Antonia SJ. Three-Year Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC-Update from PACIFIC. J Thorac Oncol. 2020 Feb;15(2):288-293. doi: 10.1016/j.jtho.2019.10.002. Epub 2019 Oct 14. PMID 31622733
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Shu CA, Gainor JF, Awad MM, Chiuzan C, Grigg CM, Pabani A, Garofano RF, Stoopler MB, Cheng SK, White A, Lanuti M, D'Ovidio F, Bacchetta M, Sonett JR, Saqi A, Rizvi NA. Neoadjuvant atezolizumab and chemotherapy in patients with resectable non-small-cell lung cancer: an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Jun;21(6):786-795. doi: 10.1016/S1470-2045(20)30140-6. Epub 2020 May 7. PMID 32386568
- [Background] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- See also: Globocan 2020 — http://gco.iarc.fr